CLINICAL TRIAL: NCT02597491
Title: Adaptive Interventions for Smoking Cessation in Lung Cancer Screening Programs
Brief Title: Program on Lung Cancer Screening and Tobacco Cessation
Acronym: PLUTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2015NTLS048
Record Dates: First submitted 2015-10-28; First posted 2015-11-05 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Smoking
Keywords: Smoking,; Smoking cessation; Sequential, multiple assignment, randomized trials (SMART); Lung cancer screening
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 4 wk assessment + TLC monthly (Active Comparator): 4 week assessment, 8 weeks of counseling, NRT, monthly follow-up (responders)
  Interventions: Behavioral: TLC monthly; Behavioral: 4 week assessment
- 4 week assessment + TLC quarterly (Active Comparator): 4 week assessment, 8 weeks of counseling, NRT, quarterly follow-up (responders)
  Interventions: Behavioral: TLC quarterly; Behavioral: 4 week assessment
- 4 week assessment +TLC + MTM (Active Comparator): 4 week assessment, 4 weeks counseling, NRT, medication management (nonresponders)
  Interventions: Behavioral: TLC monthly; Behavioral: MTM; Behavioral: 4 week assessment
- 8 week assessment + TLC monthly (Active Comparator): 8 week assessment, 8 weeks of counseling, NRT, monthly follow-up (responders)
  Interventions: Behavioral: TLC monthly; Behavioral: 8 week assessment
- 8 week assessment + TLC quarterly (Active Comparator): 8 week assessment, 8 weeks of counseling, NRT, quarterly follow-up (responders)
  Interventions: Behavioral: TLC quarterly; Behavioral: 8 week assessment
- 8 week assessment + TLC + MTM (Active Comparator): 8 week assessment, 8 weeks counseling, NRT, medication management (nonresponders)
  Interventions: Behavioral: TLC monthly; Behavioral: MTM; Behavioral: 8 week assessment

INTERVENTIONS:
Behavioral: TLC monthly — Tobacco longitudinal care monthly
  Arms: 4 week assessment +TLC + MTM; 4 wk assessment + TLC monthly; 8 week assessment + TLC + MTM; 8 week assessment + TLC monthly
Behavioral: TLC quarterly — Tobacco longitudinal care quarterly
  Arms: 4 week assessment + TLC quarterly; 8 week assessment + TLC quarterly
Behavioral: MTM — Medication management therapy
  Arms: 4 week assessment +TLC + MTM; 8 week assessment + TLC + MTM
Behavioral: 4 week assessment — 4 week assessment
  Arms: 4 week assessment + TLC quarterly; 4 week assessment +TLC + MTM; 4 wk assessment + TLC monthly
Behavioral: 8 week assessment — 8 week assessment
  Arms: 8 week assessment + TLC + MTM; 8 week assessment + TLC monthly; 8 week assessment + TLC quarterly

SUMMARY:
In this sequential, multiple assignment, randomized trial (SMART) current smokers who are eligible for lung cancer screening will be identified using the electronic medical record at the University of Minnesota and Minneapolis VA (N=1000). All participants will receive 8 weeks of evidence-based first-line smoking cessation treatment. Participants will be eligible for three potential randomizations during one year of smoking intervention: 1) to timing of identifying early response to treatment at 4 vs. 8 weeks (all participants), 2) to telephone-based tobacco longitudinal care (TLC) vs. TLC plus pharmacist-administered Medication Therapy Management (incomplete responders to first-line treatment, Primary Aim), and 3) to monthly TLC contact vs. quarterly TLC contact (complete responders to first-line treatment, Secondary Aim). The primary outcome will be 6 months of prolonged abstinence measured 18 months after the beginning of treatment.

DETAILED DESCRIPTION:
In this sequential, multiple assignment, randomized trial (SMART) current smokers who are eligible for lung cancer screening will be identified using the electronic medical record at the University of Minnesota and Minneapolis VA (N=1000). All participants will receive 8 weeks of evidence-based first-line smoking cessation treatment. Participants will be eligible for three potential randomizations during one year of smoking intervention: 1) to timing of identifying early response to treatment at 4 vs. 8 weeks (all participants), 2) to telephone-based tobacco longitudinal care (TLC) vs. TLC plus pharmacist-administered Medication Therapy Management (incomplete responders to first-line treatment, Primary Aim), and 3) to monthly TLC contact vs. quarterly TLC contact (complete responders to first-line treatment, Secondary Aim). The primary outcome will be 6 months of prolonged abstinence measured 18 months after the beginning of treatment (self-reported smoking abstinence using imputation for missing data).

ELIGIBILITY:
Inclusion Criteria:

1. scheduled or has order for low dose CT screening for lung cancer, or is eligible for screening low-dose CT
2. current daily smoker (eligible smokers will have smoked during the past 30 days and on at least 5 out of the past 7 days; individuals who have made a recent quit attempt, for example, in anticipation of their low dose CT scan for lung cancer screening, will be eligible if during the last 30 days, when they were smoking regularly, they smoked on at least 5 out of 7 days of the week).
3. 55 to 79 years old,
4. Interested in quitting and willing to choose a quit smoking date within the next 12 weeks,
5. voluntary written consent

Exclusion Criteria:

1. Unstable psychiatric disease, unless stable in treatment for 3 months (smokers on mental health medication with any changes in medication in past 3 months require study MD approval to participate) - Smokers with stable psychiatric disease will be eligible; this baseline characteristic and related symptoms will be considered in analyses,
2. No hospitalization for mental health reasons in past 3 months; No thoughts of self-harm in past 2 weeks,
3. No recent cognitive impairment (difficulties planning or organizing daily activities, such as managing finances, having trouble remembering appointments, or forgetting the correct month of the year); participants reporting recent cognitive impairment will be given the 6-item Callahan Cognitive Screener and must score at least a 5 out of 6 to participate,
4. Participating in a formal quit program (such as tobacco cessation counseling with or without use of NRT, bupropion, or varenicline; Smokers using NRT will be eligible as long as they are not using it as part of a formal quit program),
5. No phone
6. Non-English speaking
7. Current diagnosis of lung cancer

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-12; Primary Completion 2021-05-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
6 months prolonged abstinence from smoking, measured 18M after randomization | 18 months
  The primary (dichotomous) outcome for all analyses will be whether or not smokers achieve 6-month prolonged abstinence measured at 18 months after the baseline assessment. All analyses will be by intention-to-treat, and include all participants randomized to intervention, regardless of whether they are lost to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Joseph, MD, Principal Investigator — University of Minnesota

REFERENCES:
- [Background] Hughes JR, Keely JP, Niaura RS, Ossip-Klein DJ, Richmond RL, Swan GE. Measures of abstinence in clinical trials: issues and recommendations. Nicotine Tob Res. 2003 Feb;5(1):13-25. PMID 12745503
- [Derived] Fu SS, Rothman AJ, Vock DM, Lindgren BR, Almirall D, Begnaud A, Melzer AC, Schertz KL, Branson M, Haynes D, Hammett P, Joseph AM. Optimizing Longitudinal Tobacco Cessation Treatment in Lung Cancer Screening: A Sequential, Multiple Assignment, Randomized Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2329903. doi: 10.1001/jamanetworkopen.2023.29903. PMID 37615989
- [Derived] Fu SS, Rothman AJ, Vock DM, Lindgren B, Almirall D, Begnaud A, Melzer A, Schertz K, Glaeser S, Hammett P, Joseph AM. Program for lung cancer screening and tobacco cessation: Study protocol of a sequential, multiple assignment, randomized trial. Contemp Clin Trials. 2017 Sep;60:86-95. doi: 10.1016/j.cct.2017.07.002. Epub 2017 Jul 4. No abstract available. PMID 28687349

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT02597491/SAP_000.pdf